CLINICAL TRIAL: NCT06643481
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Parallel Group Study of VHB937 in Amyotrophic Lateral Sclerosis (ALS) Over 40 Weeks Followed by an Open Label Extension (ASTRALS)
Brief Title: A Clinical Trial to Learn About the Effects of VHB937 in People With Amyotrophic Lateral Sclerosis (ALS)
Acronym: ASTRALS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVHB937B12201; 2024-512536-29-00 (Other: EUCTIS)
Record Dates: First submitted 2024-09-30; First posted 2024-10-16 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis; ALS; monoclonal antibody; motor neuron disease; MND
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Intervention Model Description: Double-blind, Randomized 2:1 ratio
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded placebo for infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): I.V. infusions
  Interventions: Biological: VHB937
- Arm 2 (Placebo Comparator): I.V. infusions
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VHB937 — VHB937 solution for infusion
  Arms: Arm 1
Other: Placebo — Solution for infusion
  Arms: Arm 2

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group Phase II study to evaluate the efficacy and safety of VHB937 in participants with early-stage ALS (within 2 years of ALS symptoms onset). The study comprises a core double-blind (DB) 40-week treatment period followed by an open label extension (OLE).

DETAILED DESCRIPTION:
The main questions this trial aims to answer in comparing VHB937 to placebo are:

* How long will participants live without needing permanent help from a machine to breathe after starting the trial treatment?
* What is the change in the participant's ability to perform daily activities? This will be measured using a questionnaire called the amyotrophic lateral sclerosis functional rating scale-revised (ALSFRS-R).
* What adverse events are reported during this trial? An adverse event is any sign or symptom that participants have during a trial. Adverse events may or may not be caused by treatments in the trial. The trial doctors will check participants' ALS and general health throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years of age or older
* male or female, if of childbearing potential, strict contraception required
* have ALS confirmed by the trial doctors using different tests.
* have mild symptoms of ALS as measured by the ALSFRS-R questionnaire (total score >=30).
* have had symptoms of ALS (weakness) within 24 months of taking part in this trial.
* have not received treatment for ALS or are currently on a stable dose of an approved treatment for ALS.
* have the ability to slowly exhale a volume of air at least 60% of what is expected for the participant's sex, height and age.

Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives of screening, or within 30 days (e.g., small molecules) / or until the expected pharmacodynamic effect has returned to baseline (e.g., biologics), whichever is longer; or longer if required by local regulations.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for 24 weeks after stopping study medication.
* History or current diagnosis of cardiac conditions or ECG abnormalities indicating significant risk of safety for participants in the study.
* Clinical evidence of liver or renal disease/injury.
* Laboratory evidence of hematological abnormalities
* Presence of unstable psychiatric disease, cognitive impairment, neurological disease other than ALS, dementia or substance abuse that would impair ability of the participant to provide informed consent, in the investigator's opinion.
* Participants that reported 'yes' on any suicidal ideation section except for the "Non-Suicidal Self-Injurious Behavior" in the past 2 years as per C-SSRS.
* Presence of cancer, HIV, Hep B, Hep C, tuberculosis, uncontrolled diabetes
* History of active severe respiratory disease, including Chronic Obstructive Pulmonary Disease, interstitial lung disease or pulmonary fibrosis.
* Taking any prohibited medications

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2028-07-07 (Estimated)

PRIMARY OUTCOMES:
The composite of PAV-free survival and change in ALSFRS-R. Analysis method: Combined Assessment of Function and Survival (CAFS) | Baseline to DB Week 40
  To compare the efficacy of VHB937 vs. placebo on a composite of permanent assisted ventilation (PAV) free survival and function in DB epoch

SECONDARY OUTCOMES:
ALS Functional Rating Scale Revised (ALSFRS-R) total score | Baseline to DB Week 40 or until death or PAV (whichever occurs first) and Baseline to OLE Week 100 or until death or PAV (whichever occurs first
  To assess the efficacy of VHB937 on functional decline in DB and OLE epochs.
Slow Vital Capacity (SVC) (% of predicted normal value) | Baseline to DB Week 40 or until death or PAV (whichever occurs first) and Baseline to OLE Week 100 or until death or PAV (whichever occurs first)
  To assess the efficacy of VHB937 in delaying decline in respiratory function in DB and OLE epochs.
Ratio to baseline in Neurofilament Light (NfL) concentration in serum | DB up to Week 40; DB and OLE up to Week 100]
  To assess the effect of VHB937 on a biomarker of neurodegeneration in DB and OLE epochs.
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to end of study
  To assess the safety and tolerability of VHB937 in DB and OLE epochs.
Time to death and Time to event (death or PAV, whichever comes first). | Baseline to DB Week 40
  To assess the efficacy of VHB937 vs. placebo on survival endpoints in DB epoch.
Time to death and Time to event (death or PAV, whichever comes first) - endpoints referring to treatment policy estimand | Baseline to OLE Week 100, and Baseline to end of study
  To assess the efficacy of early vs. delayed VHB937 administration on survival endpoints (DB VHB937 followed by OLE VHB937 vs. DB placebo followed by OLE VHB937)
Patient Global Impression of change in functional ability and ALS symptom severity (PGI-C) | DB up to Week 40; DB and OLE up to Week 100
  To assess change in ALS condition in DB and OLE epochs.
Change in QoL from baseline as measured with Amyotrophic Lateral Sclerosis Assessment Questionnaire -5 (ALSAQ-5) | DB up to Week 40; DB and OLE up to Week 100
  To assess Quality of Life (QoL) with VHB937 in DB and OLE epochs.
Change in Clinician Global Impression of change in functional ability and ALS symptom severity (CGI-C) | DB up to Week 40; DB and OLE up to Week 100
  To assess change in ALS condition in DB and OLE epochs.
Change in QoL from baseline as measured with EuroQoL 5 Dimension 5 Level (EQ-5D-5L) | DB up to Week 40; DB and OLE up to Week 100
  To assess Quality of Life (QoL) with VHB937 in DB and OLE epochs.
Change in QoL from baseline as measured with 12-item Short form health survey (SF-12) | DB up to Week 40; DB and OLE up to Week 100
  To assess Quality of Life (QoL) with VHB937 in DB and OLE epochs.
Pharmacokinetics (PK) of VHB937-CMAX | Day 1 to end of study
  CMAX - The maximum concentration of VHB937 in serum
Pharmacokinetics (PK) of VHB937-TMAX | Day 1 to end of study
  TMAX - The time to reach the maximum concentration of VHB937 in serum
Pharmacokinetics (PK) of VHB937-CTROUGH | Day 1 to end of study
  CTROUGH - Minimum observed concentration of VHB937 in serum
To assess immunogenicity (IG) of VHB937 | Day 1 up to end of study
  To assess immunogenicity of Anti-VHB937 antibodies in serum
Cerebralspinal Spinal Fluid Pharmacokinetics (PK) of VHB937-CMAX | Screening to Week 12
  CMAX - The maximum concentration of VHB937 in CSF
Cerebralspinal Spinal Fluid Pharmacokinetics (PK) of VHB937-TMAX | Screening to Week 12
  TMAX - The time to reach the maximum concentration of VHB937 in CSF
Cerebralspinal Spinal Fluid Pharmacokinetics (PK) of VHB937-CTROUGH | Screening to Week 12
  CTROUGH - Minimum observed concentration of VHB937 in CSF

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (87):
- United States (24):
  - University of California San Diego, La Jolla, California
  - Loma Linda University Health, Loma Linda, California
  - Keck Medical Center USC, Los Angeles, California
  - UC San Francisco Medical Center, San Francisco, California
  - University of Miami, Miami, Florida
  - Orlando Health Clinical Trials, Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Neurology Associates P C, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Lange Neurology PC, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Atrium Health, Charlotte, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Univ of Cincinnati Medical Center, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Providence ALS Center, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - AMR Knoxville, Knoxville, Tennessee
  - Austin Neuromuscular Center, Austin, Texas
  - Nerve and Muscle Center of Texas, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
- Australia (5):
  - Novartis Investigative Site, North Ryde, New South Wales
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Cauldfield, Victoria
  - Novartis Investigative Site, Southport
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Canada (3):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Beijing, China
- Denmark (2):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Kobenhavn N V
- Novartis Investigative Site, Turku, Finland
- France (7):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Tours
- Germany (9):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Rostock, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Dublin, Ireland
- Italy (4):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Torino, TO
- Japan (5):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Ohtsu, Shiga
  - Novartis Investigative Site, Tokushima, Tokushima
  - Novartis Investigative Site, Ōta-ku, Tokyo
- Novartis Investigative Site, Utrecht, Netherlands
- Poland (4):
  - Novartis Investigative Site, Krakow, Poland
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
- South Korea (2):
  - Novartis Investigative Site, Yangsan, Gyeongsangnam-do
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago, Corunja
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Valencia
- Sweden (3):
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Sankt Gallen
- United Kingdom (4):
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Farnborough
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com